CLINICAL TRIAL: NCT04123509
Title: Non-invasive Method for Predicting the Presence of Gastroesophageal Varices in Patients With Cirrhosis: a Prospective, Single-center Trial
Brief Title: Non-invasive Method for Predicting the Presence of Gastroesophageal Varices in Patients With Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 011
Record Dates: First submitted 2019-10-07; First posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-08

CONDITIONS: Gastroesophageal Varices; Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gastroesophageal varices are a complication of portal hypertension in cirrhosis.Endoscopy is an unsatisfactory screening test.In this prospective clinical study,we will enroll patients with cirrhosis of various causes, all of whom undergo laboratory tests, elastography, and serum proteomic differential protein testing, including liver elastography (LSM) and spleen elastography (SSM). Baveno VI or expanded BavenoVI criteria are validated by comparing patients' LSM, SSM, serum differential protein, platelet count, and EGD data to evaluate the clinical value of SSM and differential proteins in excluding cirrhosis of cirrhosis.At the same time, based on SSM and serum differential protein, a new predictive model of variceal varices will be established to evaluate the diagnostic value of SSM and differential protein for esophagogastric varices, and a non-invasive method for reliably predicting and evaluating cirrhosis with esophageal varices will be found.

ELIGIBILITY:
Inclusion Criteria:

1. The age ranged from 18 to 75 years.
2. Clinical or pathological diagnosis of cirrhosis;
3. Electronic gastroscopy is planned;
4. To agree and sign the informed consent;

Exclusion Criteria:

1. Hepatocellular carcinoma or other malignant tumors have been or are currently diagnosed;
2. Orthotopic liver transplantation patients;
3. Patients who have undergone transjugular intrahepatic portosystemic shunt (TIPS),or previous surgical shunt;
4. Pregnant women;
5. Neurological or psychiatric disorders;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cirrhosis of various etiologies
Sampling Method: Probability Sample
Enrollment: 616 (Estimated)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
high-risk esophageal varices | 2 years
  Incidence of high-risk esophageal varices

SECONDARY OUTCOMES:
bleeding event happen | 1 year
  Incidence of hemorrhagic events
bleeding event happen | 2 years
  Incidence of hemorrhagic events

CONTACTS AND LOCATIONS:
Locations (1):
- Hepatology Unit, Department of Infectious Diseases, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Liu M, Zhang X, Cheng X, He Q, Zhou T, Wang H, Li B, Luo W, Li J, Li H, Lin Z, Song J, Wang W, Huang J, Ji Y, Zhou D, Xie W, Yang Q, Tu M, Luo X, Zhang X, Yan H, Chen J. Indocyanine Green Clearance Test via Pulse Dye Densitometry for Portal Hypertension Diagnosis in cACLD. Liver Int. 2025 Dec;45(12):e70425. doi: 10.1111/liv.70425. PMID 41178521
- [Derived] Sharma S, Agarwal S. Prospective validation of Baveno VI criteria in virally supressed HBV cirrhosis - more evidence is needed. J Hepatol. 2021 Mar;74(3):758-759. doi: 10.1016/j.jhep.2020.10.007. Epub 2021 Jan 19. No abstract available. PMID 33353741
- [Derived] Wang H, Wen B, Chang X, Wu Q, Wen W, Zhou F, Guo Y, Ji Y, Gu Y, Lai Q, He Q, Li J, Chen J, Hou J. Baveno VI criteria and spleen stiffness measurement rule out high-risk varices in virally suppressed HBV-related cirrhosis. J Hepatol. 2021 Mar;74(3):584-592. doi: 10.1016/j.jhep.2020.09.034. Epub 2020 Oct 8. PMID 33039403